CLINICAL TRIAL: NCT03634189
Title: Phase I, Single Center, Open-label Study of Cannabidiol in Patients With Heart Failure in AHA/ACC Stages A-C
Brief Title: Cannabidiol in Patients With Heart Failure Failure in AHA/ACC Stages A-C
Acronym: CAPITAL-AC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Cardiología y Medicina Vascular Hospital Zambrano-Hellion Tec Salud (Other)
Responsible Party: Principal Investigator, David Rodriguez, Clinical Research Coordinator, Instituto de Cardiología y Medicina Vascular Hospital Zambrano-Hellion Tec Salud
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAPITAL-AC
Record Dates: First submitted 2018-08-13; First posted 2018-08-16 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Heart Failure
Keywords: Cannabidiol; Heart Failure; AHA/ACC stage A-C
MeSH Terms: conditions — Heart Failure | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HF- ACC/AHA stage A-C + CBD (Experimental): Patients with HF stages A-C + Cannabidiol
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol — Patients with ACC/AHA stage A-C will receive 5 mg/kg to a maximum tolerated dose of 25 mg/kg PO BID of Cannabidiol

SUMMARY:
Cannabidiol in heart failure

ELIGIBILITY:
Inclusion criteria

* Men and women (women not pregnant neither in lactation period) between 30 to 75 years-old
* Patients with stage A-C of the American College of Cardiology/American Heart Association classification
* Patients with GDMT and clinical stability within four weeks
* Diagnosis of ischemic or non-ischemic dilated cardiomyopathy
* Participants should sign an informed consent form (ICF) form personally

Exclusion criteria

* Severe primary valvular cardiomyopathy or valvular prosthesis (mechanical or bio-valve)
* History of heart transplant surgery, cardiomyoplasty, left ventricular reduction surgery, valvuloplasty, implantation of a ventricle assist device and surgical cardiac congenital defect correction
* Implantable cardioverter defibrillator within the last three months
* Acute coronary syndromes that required pharmacological or mechanical reperfusion or medical treatment, within 30 days before selection
* Percutaneous coronary intervention within 30 days prior to selection
* Women who are pregnant, or of childbearing potential and are not practicing an effective means of birth control
* Untreated thyroid disease
* Hepatorenal syndrome
* History of seizures
* Hemoglobin: < 8.5 gm/dL
* WBC count lower than 3000/mm3
* Platelets: <100,000/mm
* AST or ALT >2.5 × upper limit of normal (ULN) unless related to primary disease
* Treatment with any investigational agent within 4 weeks of screening or 5 half-lives of the investigational drug (whichever is longer)
* Active cancer of any etiology
* History of psychiatric disorder (depression or PHQ-9 ≥ 10 points , bipolar syndrome, schizophrenia) or suicide attempt.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Fertile female participants not applying any approved duel anti-contraceptive method
* Inability to comply/assist with study and follow-up procedures
* Patients in cardiovascular rehabilitation programs
* Any person who is not able to give adequate ICF

Elimination criteria

* Progression of heart failure stage according to the American College of Cardiology/American Heart Association classification, since the initiation of the study.
* ALT or AST >3x normal values with a total bilirubin ≥ 2x normal value.
* Any degree of depression at any stage of the study

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related serious adverse events and events of interest as assessed by MedDRA v5.1 | 6 months
  We will assess the safety of CBD in patients with HF ACC/AHA stages A-C based on the incidence of events of interest and serious adverse events. This assessment will be performed at each on-site visit.